CLINICAL TRIAL: NCT01342757
Title: Using Proton Magnetic Resonance Spectroscopy (MRS) to Predict Response of Vorinostat Treatment in Glioblastoma
Brief Title: Magnetic Resonance Spectroscopy Imaging in Predicting Response to Vorinostat and Temozolomide in Patients With Recurrent or Progressive Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2011-02569; EMORY IRB #00044064 (Other: Emory University); WCI-44064 (Other: Winship Cancer Institute); R21CA141836 (NIH)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Adult Glioblastoma; Depression; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Depression; Brain Neoplasms | interventions — Vorinostat; Temozolomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive vorinostat once daily on days -7 to -1 (course 1 only) and days 8-14 and 22-28 and temozolomide on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients undergo magnetic resonance spectroscopic imaging at baseline and at approximately 1 and 8 weeks on treatment. Patients also undergo a survey administration of Inventory of Depression Symptomatology Self-Reported (IDS-SR) assessment at baseline and periodically during study.
  Interventions: Drug: vorinostat; Drug: temozolomide; Procedure: magnetic resonance spectroscopic imaging; Other: survey administration

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: temozolomide — Given orally
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Procedure: magnetic resonance spectroscopic imaging — Undergo MRI
  Other Names: 1H-nuclear magnetic resonance spectroscopic imaging; Proton Magnetic Resonance Spectroscopic Imaging
Other: survey administration — Ancillary studies

SUMMARY:
This clinical trial is studying magnetic resonance spectroscopy imaging in predicting response in patients to vorinostat and temozolomide in patients with recurrent, progressive, or newly diagnosed glioblastoma. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vorinostat may also help temozolomide work better by making tumor cells more sensitive to the drug. Imaging procedures, such as magnetic resonance spectroscopy imaging, may help measure the patient's response to vorinostat and temozolomide and allow doctors to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the strength of the association between magnetic resonance spectroscopy (MRS) imaging measurable biomarkers and response to vorinostat plus temozolomide.

SECONDARY OBJECTIVES:

I. To evaluate MRS-detected inositol and N-acetylaspartate (NAA) levels (at 3 tesla) as indicators of mood alterations as measured by a self-report depression survey (IDS-SR).

OUTLINE:

Patients receive vorinostat orally (PO) once daily (QD) on days -7 to -1 (course 1 only) and days 8-14 and 22-28 and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients previously treated with standard radiotherapy and temozolomide receive maintenance temozolomide PO on days 1-5.

Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicities. Patients undergo magnetic resonance spectroscopy imaging at baseline and at approximately 1 and 8 weeks on treatment. Patients also undergo an Inventory of Depression Symptomatology Self-Reported (IDS-SR) assessment at baseline and periodically during study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have 1 of the following:

  * Diagnosis of recurrent or progressive glioblastoma

    * Patients with recurrent disease may have had treatment for any number of prior relapses
  * Newly diagnosed glioblastoma and have completed radiation therapy and are receiving standard follow-up temozolomide
* Must be able to have an MRI, and have a measurable contrast-enhancing supratentorial tumor of at least 1 cm by shortest diameter
* Residual disease following resection measuring 1 cm in diameter or greater is mandated for eligibility into the study
* Patients must have a stable or progressive disease as determined by serial brain MRI using the McDonald Criteria on a scan 14 days or fewer before registration and on a stable steroid dose for 5 days
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) or thallium scanning, MR spectroscopy, or surgical documentation of disease
* White Blood Cell Count > 3,000/μL
* Absolute Neutrophil Count > 1,500/μL
* Platelet count > 100,000/μL
* Hemoglobin > 10 g/dL (transfusion allowed)
* Serum glutamate oxaloacetate transaminase < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 mg/dL
* Negative pregnancy test
* Women of childbearing potential and men must agree to use adequate barrier contraception for the duration of study participation
* Able to swallow capsules
* No patients with pacemakers, non-titanium aneurysm clips, neurostimulators, cochlear implants, non-titanium metal in ocular structures, history of being a steel worker, or other incompatible implants
* No significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* No history of any other cancer except non-melanoma skin cancer or carcinoma in-situ of the cervix, or cancer in complete remission and off all therapy for ≥ 3 years
* No active infection or serious intercurrent medical illness
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat (SAHA) or other agents used in this study
* No prolonged corrected QT interval waves on baseline EKG
* No other anticancer therapy (including chemotherapy, radiation, hormonal treatment, or immunotherapy) of any kind is permitted during the study period
* At least 3 weeks since prior radiotherapy
* Patients must have recovered from the toxic effects of prior therapy, including surgery
* At least 28 days since any prior investigational agent or prior cytotoxic therapy
* At least 23 days since prior temozolomide
* At least 14 days since prior vincristine (42 days for nitrosourea)
* At least 21 days since prior procarbazine
* At least 7 days since prior non-cytotoxic agents (e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc.)
* At least 2 weeks since prior valproic acid (or another histone deacetylase inhibitor)
* No other concurrent investigational agents

Exclusion Criteria:

* Diagnostic and Statistical Manual-IV Axis I or II diagnosis (as determined by PI), exclusive of nicotine dependence.
* Pregnant.
* Contraindications to MRI: pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
* Active medical or neurological disorder.
* History of alcohol or drug dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olson, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Shim H, Wei L, Holder CA, Guo Y, Hu XP, Miller AH, Olson JJ. Use of high-resolution volumetric MR spectroscopic imaging in assessing treatment response of glioblastoma to an HDAC inhibitor. AJR Am J Roentgenol. 2014 Aug;203(2):W158-65. doi: 10.2214/AJR.14.12518. PMID 25055291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment closed
Pre-assignment Details: No events requiring changes in approach or enrollment criteria
Groups:
- Vorinostat and Temozolomide: Patients receive vorinostat orally (PO) once daily (QD) on days -7 to -1 (course 1 only) and days 8-14 and 22-28 and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients previously treated with standard radiotherapy and temozolomide receive maintenance temozolomide PO on days 1-5.
  Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicities. Patients undergo magnetic resonance spectroscopy imaging at baseline and at approximately 1 and 8 weeks on treatment. Patients also undergo an Inventory of Depression Symptomatology Self-Reported (IDS-SR) assessment at baseline and periodically during study.
Period: Overall Study
Arm/Group | Vorinostat and Temozolomide
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive vorinostat orally (PO) once daily (QD) on days -7 to -1 (course 1 only) and days 8-14 and 22-28 and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients previously treated with standard radiotherapy and temozolomide receive maintenance temozolomide PO on days 1-5.
  Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicities. Patients undergo magnetic resonance spectroscopy imaging at baseline and at approximately 1 and 8 weeks on treatment. Patients also undergo an Inventory of Depression Symptomatology Self-Reported (IDS-SR) assessment at baseline and periodically during study.
Arm/Group | Arm I
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Magnetic Resonance Spectroscopy (MRS) Response to Initial Vorinostat by MRI and MRS Scans as Determined by Spectroscopic Index
Description: Changes in magnetic resonance spectroscopic imaging signal and semiquantitative analysis of inositol, choline, lactate, and N-acetylaspartate signal are measured. The values for each of these metabolites are normalized to baseline at one and nine weeks. The values of all the metabolites at one week are added and this is the magnetic resonance spectroscopic index for one week. This is done again at nine weeks. The number is unitless and there is no range limit. Positive values represent normalization of tumor metabolism and negative values suggest no improvement or worsening of metabolic character.
Time Frame: 9 weeks
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 12
participants | 0

2. Primary Outcome: Proportion of Patients Who Experience Metabolic Restoration Between the Responders and Non-responder Groups by MRS Scans
Description: Baseline MRS was performed 1-3 days before initiation of treatment. Follow-up MRS studies were performed at day 7. A standard quadrature head coil was used to collect MR data. A responder was defined as stable disease: determined in glioblastoma to be between a 25% volume increase and 50% volume decrease compared to baseline imaging at the therapy initiation at the 2 month follow-up visit. The spectroscopic restoration index was calculated (ΔN-acetyl aspartate + Δcreatine + Δmyo-inositol - Δcholine - Δ(lactate / lipids)).
Time Frame: After 1 week
Population: In five of the twelve cases spectroscopic indices could not be calculated because the tumor volume was outside of reliably measured voxels. These were primarily accounted for by tumor closeness to the skull or the small size of residual tumor.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 7
Participants
  Metabolic Responders SRI Greater than 0 | 3
  Metabolic Responders SRI 0 or Less | 0
  Metabolic Non-Responders SRI Greater than 0 | 0
  Metabolic Non-Responders SRI 0 or Less | 4

3. Primary Outcome: Measurable Change on Magnetic Resonance Spectroscopy Imaging After Vorinostat Administration
Description: Changes in magnetic resonance spectroscopic imaging signal and semiquantitative analysis of inositol, choline, lactate, and N-acetyl aspartate (NAA) signal are measured. The values for each of these metabolites are normalized to baseline at one and nine weeks. The values of all the metabolites at one week are added and this is the magnetic resonance spectroscopic index for one week. This is done again at nine weeks. The number is unitless and there is no range limit. Positive values represent normalization of tumor metabolism and negative values suggest no improvement or worsening of metabolic character.
Time Frame: 9 weeks
Population: Patients collected until measurable spectroscopic indexes were available in at least three cases with metabolic response and three without metabolic response
Measure: Mean (Standard Deviation); unit: Spectroscopic index
Arm/Group | Arm I
Number analyzed (Participants) | 12
Spectroscopic index | 0 (1.4)

4. Secondary Outcome: Mean Change in Metabolite Levels
Description: Baseline MRS was performed 1-3 days before initiation of treatment. Follow-up MRS studies were performed at day 7. A standard quadrature head coil was used to collect MR data. The change of metabolite level in choline (Cho) and N-acetyl aspartate (NAA) were calculated in ratio by (metabolite after treatment / metabolite before treatment - 1). The reported ratios represent the Cho-to-NAA ratio at day 7 compared with day 0.
Time Frame: Baseline to 1 week
Measure: Mean (Full Range); unit: Cho/NAA Ratios
Arm/Group | Arm I
Number analyzed (Participants) | 7
Cho/NAA Ratios
  Metabolic Responders | -0.15 [-0.32 to -0.04]
  Metabolic Non-Responders | 0.29 [0 to 0.94]

ADVERSE EVENTS:
Time Frame: Until tumor progression by imaging
Description: Clinic visits, drug diary and patient reporting
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=12)
Thromboembolism (Vascular disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=12)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Edema in Limbs and Hands (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Skin infection-scalp (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4)
Bruising (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALT increased (Metabolism and nutrition disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Creatinine Increased (Renal and urinary disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Intracranial Hemorrhage (Nervous system disorders) | 2 (2)
Weight Loss (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
AST elevation (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Weakness, left sided (Nervous system disorders) | 1 (1)
Prolonged APTT (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Cognitive Disturbances (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Gastoesophageal Reflux disease (Gastrointestinal disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
In five of the twelve cases spectroscopic indices could not be calculated because the tumor volume was outside of reliably measured voxels. These were primarily accounted for by tumor closeness to the skull or the small size of residual tumor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less